CLINICAL TRIAL: NCT02778750
Title: Evaluation Of The Pan-microbiome and Host Immune Response in Cystic Fibrosis (CF)
Brief Title: Evaluation Of The Pan-microbiome and Host Immune Response in CF
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01692
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stable Group
  Interventions: Procedure: Two-Bronchoscope Technique
- Rapid Decliner Group
  Interventions: Procedure: Two-Bronchoscope Technique

INTERVENTIONS:
Procedure: Two-Bronchoscope Technique — Used to validate the use of sputum to sample the lower airway microbiome

SUMMARY:
Investigators will examine temporal and regional dynamic changes in the microbiome of Cystic Fibrosis patients to explore microbiome features that are associated with an inflammatory phenotype. Investigators hypothesize that temporal and spatial differences in lung microbiome are associated with host inflammatory responses.

While chronic and polymicrobial airway colonization are commonly recognized in cystic fibrosis (CF), it is unclear what factors of the microbial environment lead to infection with pathogenic microorganism. This is a multi center, longitudinal cohort of adult Cystic Fibrosis subjects recruit4ed from NYU and Columbia to understand how changes in the airway microbiome may affect the host inflammatory responses in Cystic Fibrosis (CF). There will be three approaches to understanding inflammatory responses; 1) a longitudinal assessment of temporal changes in the microbiome over a 6-month period of clinical stability; 2) comparison of the regional differences in airway microbiome between lung segments with more versus less disease; 3) evaluation of functional aspects of the lung microbiome.

ELIGIBILITY:
Inclusion Criteria:

* CF diagnosis
* able to produce sputum
* no recent (one month) exacerbation defined as physician treatment with antibiotics for ≥ 7days
* FEV1 ≥ 30% of predicted.

Exclusion Criteria:

* Initiation of any new chronic therapy (e.g., ibuprofen, aerosolized rhDNase, hypertonic saline, azithromycin, tobramycin inhalation solution, aztreonam inhalation solution, ivacaftor) within 8 weeks prior to enrolment
* introduction of vitamins or proton pump inhibitors within 8 weeks prior to enrolment
* use of new investigational therapy within 4 weeks
* current smoker; use of oral corticosteroids
* Initiation of treatment or change in regimen for allergic bronchopulmonary aspergillosis or nontuberculous mycobacteria within 8 weeks.
* liver enzymes > 3 times the upper limit
* pregnancy

Additional Exclusion Criteria for Bronchoscopy Subgroup (Aims 2 and 3):

* FEV1 < 50% of predicted.
* Significant cardiovascular disease defined as abnormal EKG, known or suspected coronary artery disease or congestive heart failure.
* Significant renal disease (Creatinine Clearance < 30%).
* Severe malnutrition (BMI <18kg/m2)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter study to create a longitudinal cohort of adult CF subjects recruited from NYU and Columbia. A subgroup of subjects will be selected for a more invasive assessment of the lung microbiome with research bronchoscopy.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Changes in Oral Inflammatory markers | Baseline, 6 Months
Changes in Sputum Inflammatory Markers measured using research bronchoscopy | Baseline, 6 Months
Changes in Gut Microbiome | Baseline, 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Segal, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States